CLINICAL TRIAL: NCT02753023
Title: Registry Of Acute meDical Emergencies in Brazil - ROAD-Brazil
Brief Title: Registry Of Acute meDical Emergencies in Brazil
Acronym: ROAD-Brazil
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PSInCor-ROAD-Brazil
Record Dates: First submitted 2016-04-26; First posted 2016-04-27 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndromes; Heart Failure; Pulmonary Edema; Aortic Aneurysm, Familial Thoracic 1; Chest Pain; Pulmonary Embolism; Syncope
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Pulmonary Edema; Aortic Aneurysm, Familial Thoracic 1; Chest Pain; Pulmonary Embolism; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- acute coronary syndromes: No intervention related
  Interventions: Other: no intervention
- acute decompensated heart failure: No intervention related
  Interventions: Other: no intervention
- warfarin intoxication: No intervention related
  Interventions: Other: no intervention
- acute pulmonary edema: No intervention related
  Interventions: Other: no intervention
- acute aortic dissection: No intervention related
  Interventions: Other: no intervention
- chest pain: No intervention related
  Interventions: Other: no intervention
- pulmonary embolism: No intervention related
  Interventions: Other: no intervention
- syncope: No intervention related
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention related

SUMMARY:
Critical patients in emergency room are seriously situations that need quickly diagnosis and treatment. Different predictors of prognosis can be related with mortality and morbidity in-hospital and in long-term. In Brazil, this kind of registry is not available. The aim of the study is analysis and report data about critical patients in Emergency Departments over all country, showing demographic, clinical and prognosis data about that in Brazil.

DETAILED DESCRIPTION:
This will be a prospective and multicentric data-bank registry. Initially, all patients with acute coronary syndromes (ACS), acute decompensated heart failure (ADHF), warfarin intoxication, acute pulmonary edema, acute aortic dissection, chest pain, pulmonary embolism and syncope will be included. There will be not exclusion criteria. The inclusion criteria will be followed by definition of each illness described in recent guidelines. Investigators estimated annually over than 500 cases with ACS/chest pain, 300 cases of ADHF, 200 cases of aortic dissection, 200 of pulmonary embolism, 200 cases of warfarin intoxication, 100 cases of syncope and 150 of acute pulmonary edema. Clinical data, electrocardiographic and echocardiographic findings, laboratory results and prognosis will be related. Routine of treatment will be defined by each center. The analysis includes minimum, medium and maximum values. Variables will be adjusted according with each diagnosis and all data will be included using the REDCap digital data entry. Probabilities will be determined by logistic regression and will be considered significate when p < 0.005. Prospectively, investigators will use the Cox model to calculate associations.

ELIGIBILITY:
Inclusion Criteria:

* all patients with:
* acute coronary syndromes (ACS) or,
* acute decompensated heart failure (ADHF) or,
* warfarin intoxication or,
* acute pulmonary edema or,
* acute aortic dissection or,
* chest pain or,
* pulmonary embolism or
* syncope.

Exclusion Criteria:

-There will be not exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency unit patients
Sampling Method: Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
mortality | 6 months

SECONDARY OUTCOMES:
mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Pronto Socorro - Hospital Metropolitano, Vitória, Espírito Santo
  - Unidade Coronariana do Hospital Estadual Mario Covas, Santo André, São Paulo
  - Hospital Unimed Sorocaba, Sorocaba, São Paulo
  - Instituto do Coração - HMFMUSP, São Paulo
  - Pronto Atendimento - Hospital Alemão Oswaldo Cruz, São Paulo
  - Pronto Socorro - Hospital TotalCor, São Paulo

IPD SHARING:
Plan to Share IPD: No